CLINICAL TRIAL: NCT02120859
Title: Fractional Flow Reserve - Guided Elective Coronary Angioplasty Using Paclitaxel - Eluting Balloons With Provisional Stent Implantation: A Phase 4 Feasibility Study With 6-Month Follow-up by Optical Coherence Tomography
Brief Title: Optical Coherence Tomography to Investigate FFR-Guided DEB-only Elective Coronary Angioplasty
Acronym: OCTOPUS-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Responsible Party: Principal Investigator, Tudor C. Poerner, MD, PD Dr. med. Tudor C. Poerner, University of Jena
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKJ-TCP-2
Record Dates: First submitted 2014-04-19; First posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Stable Angina; Coronary Stenosis
Keywords: PCI; Drug-eluting balloon (DEB); Fractional flow reserve (FFR)
MeSH Terms: conditions — Angina, Stable; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FFR - guided DEB angioplasty (Experimental): DEB-only angioplasty is attempted in all patients. At baseline, quantitative coronary angiography (QCA) and fractional flow reserve (FFR) using an intracoronary standard bolus of adenosine are performed. If FFR at baseline is greater than 0.8, PCI is deferred, otherwise predilation with a non-coated balloon is performed. In case of severe recoil (> 50% residual stenosis) or flow-limiting dissection the procedure is deemed not suitable for DEB-only angioplasty and stent implantation is performed at the discretion of the operator. In all other cases, the lesion is treated using a Sequent Please® paclitaxel-eluting balloon (DEB). QCA and FFR measurements are repeated and the result is considered satisfactory if there is no flow-limiting dissection, residual stenosis < 40% and FFR > 0.8.
  Interventions: Device: FFR - guided DEB angioplasty
- DEB angioplasty with provisional bare metal stenting (Other): In case of suboptimal results after the FFR-guided DEB angioplasty described above, a bare metal stent is implanted inside the segment previously treated by DEB.
  Interventions: Device: FFR - guided DEB angioplasty; Device: Provisional bare metal stenting

INTERVENTIONS:
Device: FFR - guided DEB angioplasty — DEB-only angioplasty is attempted in all patients. At baseline, quantitative coronary angiography (QCA) and fractional flow reserve (FFR) using an intracoronary standard bolus of adenosine are performed. If FFR at baseline is greater than 0.8, PCI is deferred, otherwise predilation with a non-coated balloon is performed. In case of severe recoil (> 50% residual stenosis) or flow-limiting dissection the procedure is deemed not suitable for DEB-only angioplasty and stent implantation is performed at the discretion of the operator. In all other cases, the lesion is treated using a Sequent Please® paclitaxel-eluting balloon (DEB). QCA and FFR measurements are repeated and the result is considered satisfactory if there is no flow-limiting dissection, residual stenosis < 40% and FFR > 0.8.
  Other Names: Sequent Please® paclitaxel-eluting balloon (DEB)
Device: Provisional bare metal stenting — In case of suboptimal results after the FFR-guided DEB angioplasty described above, a bare metal stent is implanted inside the segment previously treated by DEB.
  Other Names: Coroflex Blue® bare metal stent (BMS)
  Arms: DEB angioplasty with provisional bare metal stenting

SUMMARY:
We aimed to evaluate feasibility and the 6-month angiographic and OCT results of FFR - guided use of paclitaxel-eluting balloons (Sequent Please™, B Braun) with provisional bare metal stenting for elective PCI of de novo coronary lesions.

DETAILED DESCRIPTION:
Restenosis rates after plain-old balloon angioplasty (POBA) are with 30-50 % very high. Therefore, this interventional concept is of limited use today. However, dual antiplatelet therapy (DAPT) is not necessary after POBA. Contrary, 3rd generation drug-eluting stents (DES) proved to be very effective showing delayed restenosis only in 5-15%, but require DAPT for at least 6 months. Drug-eluting balloons (DEB) might be a promising trade-off between POBA and DES, since they effectively inhibit neointimal proliferation despite minimal duration of DAPT. However, there is still very limited data on this interventional strategy. Thus, we aimed to investigate feasibility of fractional flow reserve (FFR) - guided use of paclitaxel-eluting balloons (Sequent Please™, B Braun) with provisional bare metal stenting for elective PCI of de novo coronary lesions, evaluating the 6-month outcomes by angiography and optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* Indication for elective PCI according to the guidelines of European Society of Cardiology, American Heart Association and American College of Cardiology
* Age > 18 years, written consent
* Native de novo coronary lesion suitable for angioplasty and OCT imaging

Exclusion Criteria:

* Pregnancy and breast feeding mother
* Co-morbidity with an estimated life expectancy of < 50 % at 1 year
* Scheduled major surgery in the next 6 months
* Not able to give informed written consent or non-compliance
* Participation in other PCI trial
* Acute coronary syndromes and cardiogenic shock
* Known allergy to aspirin, thienopyridines or against taxol derivates
* Culprit lesion within the proximal 10 mm of the right or left coronary artery
* Saphenous vein grafts
* Estimated lesion length > 30 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Late lumen loss | 6 months
  Late lumen loss (LLL, expressed in mm) measured within the treated segment by quantitative coronary angiography (QCA) as the difference between minimal luminal diameter (MLD) at the end of the interventional procedure and MLD at 6-month follow-up

SECONDARY OUTCOMES:
Vessel remodeling assessed by optical coherence tomography | 6 months
  Lumen and vessel measurements, neointimal proliferation, plaque composition and dissection healing within the treated vessel segment at 6 months assessed by optical coherence tomography (OCT) with 3D-reconstruction
Net lumen gain | 6 months
  Net lumen gain (NLG, expressed in mm) measured by quantitative coronary angiography (QCA) as the difference between minimal luminal diameter within the treated segment (MLD) at 6-month follow-up and MLD at the lesion site at baseline
Need for revascularization of the treated vessel segment | 6 months
  Need for revascularization of the treated vessel segment (target lesion revascularization, TLR) driven either clinically or after 6-month angiographic follow-up

OTHER OUTCOMES:
Cardiac death or acute myocardial infarction due to target vessel failure | 6 month
  Cardiac death or acute myocardial infarction occurring in the presence of occlusion or severe flow limitation of the treated vessel

CONTACTS AND LOCATIONS:
Overall Officials: Tudor C Poerner, MD, Study Director — University Hospital of Jena, Heart Center, Cardiology Division; Hans R Figulla, MD, Study Chair — University Hospital of Jena, Heart Center, Cardiology Divisio
Locations (1):
- University Hospital of Jena, Heart Center, Division of Cardiology, Jena, Germany

REFERENCES:
- [Derived] Poerner TC, Duderstadt C, Goebel B, Kretzschmar D, Figulla HR, Otto S. Fractional flow reserve-guided coronary angioplasty using paclitaxel-coated balloons without stent implantation: feasibility, safety and 6-month results by angiography and optical coherence tomography. Clin Res Cardiol. 2017 Jan;106(1):18-27. doi: 10.1007/s00392-016-1019-4. Epub 2016 Jul 5. PMID 27379610